CLINICAL TRIAL: NCT06076824
Title: Glucocorticoid Treatment in Patients Undergoing TAVR to Reduce the Incidence of Atrioventricular Block and Pacemaker Implantation
Brief Title: Glucocorticoid Treatment in Transaortic Valve Replacement to Reduce the Incidence of Conduction Disturbances (GLUCO-TAVR).
Acronym: GLUCO-TAVR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General Universitario de Alicante (Other)
Responsible Party: Principal Investigator, Juan Miguel Ruiz Nodar, Head of the department of Interventional Cardiology and Principal Investigator, Hospital General Universitario de Alicante
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-116
Record Dates: First submitted 2023-09-26; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Heart Block; Aortic Stenosis; Bundle-Branch Block
Keywords: Transcatheter Aortic Valve Replacement; Glucocorticoids; Inflammation; Conduction disturbances; Heart block
MeSH Terms: conditions — Heart Block; Aortic Valve Stenosis; Bundle-Branch Block; Inflammation | interventions — Methylprednisolone; Saline Solution

STUDY DESIGN:
Intervention Model Description: Phase IV, single-center, randomized, controlled, and open label clinical trial (with blinded outcomes assessor).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Glucocorticoid treatment) (Experimental)
  Interventions: Drug: Methylprednisolone
- Control group (Placebo Comparator): Saline solution (0.9%)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Methylprednisolone — The intervention group will recieve 7 mg/kg/day (or a maximum of 500 mg/day) of intravenous Methylprednisolone an hour before TAVR followed by 15 mg / 12h of Prednisone during 5 days after the intervention (starting 24h after the administration of Methylprednisolone).
  Arms: Intervention group (Glucocorticoid treatment)
Other: Placebo — Saline solution
  Other Names: Saline solution
  Arms: Control group

SUMMARY:
The goal of this phase IV, randomized, controlled and open-label study is to assess the efficacy of peri-procedure glucocorticoid treatment in the prevention of conduction abnormalities and the need for pacemaker implantation in patients undergoing transaortic valve replacement compared to placebo. Participants randomized to the intervention group will receive a single dose of intravenous Methylprednisolone 7 mg/kg/day on the day of the procedure (1 hour before), followed by 15 mg/12 hours of daily Prednisone for 5 days.

The primary endpoint is a composite of permanent pacemaker implantation and the occurrence of new conduction abnormalities (any-degree AV block, bundle branch block, or non-specific intraventricular conduction disorder) at discharge, at 30 days and 1 year.

DETAILED DESCRIPTION:
Aortic stenosis is the most common valvular heart disease in Europe, and its prevalence is expected to increase in the coming years. The definitive treatment is aortic valve replacement through surgery or transcatheter aortic valve implantation (TAVR). TAVR emerged as an alternative to surgery for high-surgical-risk patients, but it has also proven effective in intermediate or low surgical-risk cases, leading to an expected rise in procedures in the near future. The most frequent complication is atrioventricular block (AVB) and permanent pacemaker implantation (PPM), which has been associated with increased morbidity, hospital stay, and healthcare costs. However, it has been suggested that post-TAVR AVB may be a transient process due to the inflammatory response triggered by the procedure. Treating this inflammation could reduce the risk of AVB after TAVR, potentially benefiting both the economy and patient outcomes.

The investigators propose a phase IV, single-center, randomized, controlled trial with an unmasked evaluator to evaluate the effect of glucocorticoids on the prevention of conduction abnormalities and PPM in TAVR patients. 100 patients will be recruited (50 in the control group and 50 in the intervention group) undergoing TAVR at the General University Hospital Dr. Balmis in Alicante, excluding those with prior PPM, chronic corticosteroid treatment, or any contraindications to these drugs. The intervention group will receive a single dose of intravenous Methylprednisolone 7 mg/kg/day on the day of the procedure (1 hour before), followed by 15 mg/12 hours of daily Prednisone for 5 days. The inflammatory response and the occurrence of conduction abnormalities will be assessed through blood tests, electrocardiograms, and echocardiography. Data will be processed using IBM-SPSS version 25.0 statistical software.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for TAVR implantation according to current European Society of Cardiology guidelines: patients with severe symptomatic aortic stenosis that are > 75 years old or have a high surgical risk.

Exclusion Criteria:

* Patients with a prior pacemaker.
* Patients with contraindications for the use of glucocorticoids including immunosuppression, active or latent infection, documented hypersensitivity or allergy, insulin-dependent diabetes mellitus, glaucoma (both closed-angle and open-angle), recent intestinal perforation, or acute heart failure.
* Patients on prior chronic treatment with glucocorticoids (both oral, inhaled, or intravenous, but topical and ophthalmic administration is allowed).
* Access for TAVR implantation other than femoral (for example, transapical).
* Patients on medication that may interact with glucocorticoids.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-12 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients that requiere pacemaker implantation and/or who develop new conduction abnormalities (AV block, bundle branch block, and/or non-specific intraventricular conduction disorder). | One week, 30 days, and 1 year after admission

SECONDARY OUTCOMES:
All-cause mortality | One week, 30 days, and 1 year after admission
Incidence of strokes (ischemic, hemorrhagic, and/or other unspecified types) | One week, 30 days, and 1 year after admission
Incidence of bleeding events requiring transfusion or life-threatening bleeding (BARC 3 or 5) | One week after admission
Incidence of major vascular complications | One week and 30 days after admission
Length of hospital stay | One week after admission
Rate of adverse events related to the use of glucocorticoids | One week and 30 days after admission
  Number of episodes of hyperglycemia, hypertensive crisis, acute decompensated heart failure and local and systemic infections
Pacemaker dependency in patients who have undergone pacemaker implantation | At 30 days and one year after admission
  Percentage of stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- General University Hospital of Alicante, Alicante, Spain